CLINICAL TRIAL: NCT03304912
Title: Packaging Pre-Exposure Prophylaxis (PrEP) to Prevent HIV Transmission Among Women Who Inject Drugs
Brief Title: Packaging PrEP to Prevent HIV Among WWID
Status: Completed | Type: Observational
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Alexis Roth, Assistant Professor, Drexel University
Other Study IDs: 1R21DA043417-01A1 (NIH)
Record Dates: First submitted 2017-09-29; First posted 2017-10-09 (Actual); Results first posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-06

CONDITIONS: HIV/AIDS
Keywords: Pre-Exposure Prophylaxis; Injection Drug Use
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women who inject drugs who are eligible for PrEP: Women who inject drugs who are eligible for PrEP are provided PrEP Education and option to accept a PrEP prescription.
  Interventions: Behavioral: PrEP Education and option to accept a PrEP prescription

INTERVENTIONS:
Behavioral: PrEP Education and option to accept a PrEP prescription — Participants will receive educational information about PrEP, be offered a PrEP prescription, and those who choose to initiated PrEP will be monitored for side-effects and adherence at their follow-up visit. There is no group assignment within this study and WWID do not have to choose to initiate PrEP. Rather, the goal of this study is to understand factors that impact PrEP initiation (and engagement in the PrEP care continuum).

SUMMARY:
Evidence suggests women who inject drugs (WWID) are disproportionately vulnerable to HIV. If HIV incidence continues unchecked, 1 in 23 WWID in the United States will acquire HIV. This observational study will evaluate a novel approach for the delivery of pre-exposure prophylaxis (PrEP) care: pairing PrEP with community-based syringe exchange program (SEP) services. The rationale is that (1) SEPs may currently provide prescription medications and long-term monitoring for other conditions such as buprenorphine for opioid dependence, so providing PrEP care is a natural extension of what is already being done successfully; (2) SEPs are a viable access point for many HIV-uninfected WWID who would be considered eligible for PrEP under current clinical guidelines; and (3) PrEP interventions, delivered in settings already utilized and trusted by WWID, will increase uptake, adherence and retention in PrEP. We will enroll a cohort of 125 women and follow-them over six months. At their first study visit, they will educated about and offered a prescription for PrEP. Those who indicate an interest in PrEP will be able to return to the SEP one week later to obtain a paper PrEP prescription or medication. All participants will be followed for six months using qualitative interviews and surveys to understand facilitators and barriers to PrEP uptake and engagement over time. In addition, we will collect urine and test it to detect the level of drug concentration among women who initiate PrEP. This will allow us to know whether their level of adherence translated to prevention effective drug levels.

DETAILED DESCRIPTION:
This prospective mixed methods study will be initiated within the largest SEP in the mid-Atlantic region. Over six months, we will use semi-structured and in-depth interviews based on the Behavioral Model for Vulnerable Populations, and drug-level monitoring for emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) adherence, to address the following specific aims: (1) Describe WWID's engagement in the PrEP care continuum (focusing on critical moments when women could disengage or need additional support to remain in care). (2) Identify factors from the Behavioral Model for Vulnerable Populations that are associated with WWID's engagement in the PrEP care continuum. (3) Explore how and why model factors are associated with WWID's decisions and ability to engage in PrEP care. A paired model of PrEP and SEP services has yet to be tested.

ELIGIBILITY:
Inclusion Criteria:

* HIV sero-negative
* Females
* Age ≥18 years
* Reporting non-prescription injection drug use and any of the following:

  1. Syringe sharing
  2. Injecting drugs with a HIV-positive partner
  3. Recent opioid agonist treatment but still injecting drugs
  4. Sex exchange
  5. Inconsistent condom use
  6. Recent bacterial sexually transmitted infection (STI)
  7. and/or sex with a HIV-positive partner

Exclusion Criteria:

* HIV seropositivity
* Currently taking PrEP
* Pregnant, breastfeeding or trying to become pregnant
* Previous enrollment in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample to be recruited from a syringe exchange program.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis M Roth, PhD, MPH, Principal Investigator — Drexel University
Locations (1):
- Drexel University Dornsife School of Public Health, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
N/A, Individual Participant Data (IPD) will not be shared.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 participants were withdrawn following enrollment because we were unable to draw blood in order to be able to prescribe PrEP medication.
Groups:
- Women Who Inject Drugs (WWID) Who Are Eligible for Pre-exposure Prophylaxis (PrEP): The cohort will be comprised of WWID who are eligible for PrEP.
  PrEP Education and option to accept a PrEP prescription: Participants will receive educational information about PrEP, be offered a PrEP prescription, and those who choose to initiated PrEP will be monitored for side-effects and adherence at their follow-up visit. There is no group assignment within this study and WWID do not have to choose to initiate PrEP. Rather, the goal of this study is to understand factors that impact PrEP initiation (and engagement in the PrEP care continuum).
Period: Overall Study
Arm/Group | Women Who Inject Drugs (WWID) Who Are Eligible for Pre-exposure Prophylaxis (PrEP)
Started | 95
Completed | 42
Not Completed | 53

BASELINE CHARACTERISTICS:
Groups:
- PrEP Education and Option to Accept a PrEP Prescription: Participants will receive educational information about PrEP, be offered a PrEP prescription, and those who choose to initiated PrEP will be monitored for side-effects and adherence at their follow-up visit. There is no group assignment within this study and WWID do not have to choose to initiate PrEP.
Arm/Group | PrEP Education and Option to Accept a PrEP Prescription
Number analyzed (Participants) | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 95
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 84
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 66
  More than one race | 4
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 95

OUTCOME MEASURES:

1. Primary Outcome: PrEP Uptake at Week 1
Description: Number of WWID accepting a paper Truvada prescription to fill at their preferred pharmacy or obtaining Truvada from the SSP among those who returned to care as verified in electronic medical records.
Time Frame: 1 week
Population: Of the 95 WWID who were offered a PrEP prescription, 89 women returned at week 1.
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP Education and Option to Accept a PrEP Prescription
Number analyzed (Participants) | 89
Participants | 63

2. Secondary Outcome: PrEP Uptake at Week 12
Description: as for outcome 1
Time Frame: 12 weeks
Population: Number of WWID returning to care at week 12.
Measure: Count of Participants; unit: Participants
Groups:
- WWID Who Are Eligible for PrEP: The cohort will be comprised of women who inject drugs who are eligible for PrEP.
  PrEP Education and option to accept a PrEP prescription: Participants will receive educational information about PrEP, be offered a PrEP prescription, and those who choose to initiated PrEP will be monitored for side-effects and adherence at their follow-up visit. There is no group assignment within this study and WWID do not have to choose to initiate PrEP. Rather, the goal of this study is to understand factors that impact PrEP initiation (and engagement in the PrEP care continuum).
Arm/Group | WWID Who Are Eligible for PrEP
Number analyzed (Participants) | 59
Participants | 48

3. Secondary Outcome: PrEP Adherence Based on Urinalysis at 12 Weeks
Description: Protection effective emtricitabine (FTC) concentration (>1000 ng/ml) in urine. Analyzed only among women with available urine-analysis data that self-reported PrEP use at 12 weeks
Time Frame: 12 weeks
Population: Women with available urine-analysis data that self-reported PrEP use at 3-months
Measure: Count of Participants; unit: Participants
Arm/Group | WWID Who Are Eligible for PrEP
Number analyzed (Participants) | 20
Participants | 1

4. Secondary Outcome: PrEP Adherence Based on Self-report at 12 Weeks
Description: Self-reported adherence was assessed with a single item administered on a computer assisted self-interview. The item, "How many PrEP pills have you missed in the past 7 days?," had numerical response options ranging from zero to seven. Responses were recoded into: took zero doses within 7 days (operationalized as non-adherent), took 1-5 doses within 7 days defined as inconsistent operationalized), and took 6-7 doses within 7 days (operationalized as consistent adherence).
Time Frame: 12 weeks
Population: Number of women responding to adherence measure on survey
Measure: Count of Participants; unit: Participants
Arm/Group | WWID Who Are Eligible for PrEP
Number analyzed (Participants) | 51
Participants
  Non-adherence | 18
  Inconsistent-adherence | 9
  Adherence | 24

5. Secondary Outcome: PrEP Uptake at Week 24
Description: as for outcome 1
Time Frame: 24 weeks
Population: Number of women returning to care at week 24
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP Education and Option to Accept a PrEP Prescription
Number analyzed (Participants) | 42
Participants | 25

ADVERSE EVENTS:
Time Frame: 6 months
Description: The definitions of adverse events and serious adverse events did not differ from the clinicaltrials.gov.
Groups:
- Women Who Inject Drugs (WWID) Who Are Eligible for PrEP.: The cohort will be comprised of women who inject drugs who are eligible for PrEP.
  PrEP Education and option to accept a PrEP prescription: Participants will receive educational information about PrEP, be offered a PrEP prescription, and those who choose to initiated PrEP will be monitored for side-effects and adherence at their follow-up visit. There is no group assignment within this study and WWID do not have to choose to initiate PrEP. Rather, the goal of this study is to understand factors that impact PrEP initiation (and engagement in the PrEP care continuum).
Arm/Group | Women Who Inject Drugs (WWID) Who Are Eligible for PrEP.
All-Cause Mortality (participants affected / at risk) | 1/95
Serious Adverse Events (participants affected / at risk) | 3/95
Other Adverse Events (participants affected / at risk) | 9/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women Who Inject Drugs (WWID) Who Are Eligible for PrEP. (N=95)
Hospitalization (General disorders) | 3 (3) — Study participant is hospitalized whether it's determined to be related to study involvement or not.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women Who Inject Drugs (WWID) Who Are Eligible for PrEP. (N=95)
Victimization (General disorders) | 9 (9) — Study participant reports they have been physically assaulted in some manner during the course of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT03304912/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT03304912/ICF_001.pdf